CLINICAL TRIAL: NCT07382518
Title: A Study on the Effects of Different Types of Self-Talk on Strikers in Soccer
Brief Title: Effects of Motivational and Instructional Self-Talk on Performance and Stress in Soccer Forwards
Acronym: STF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Sport University (Other)
Responsible Party: Principal Investigator, Yue Dou, Graduate Student, Beijing Sport University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2025556H
Record Dates: First submitted 2026-01-27; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2026-01

CONDITIONS: Psychological Self-talk Interventions in Soccer Performance
Keywords: Self-talk; Soccer; Psychological intervention; Athletic performance; Stress regulation

STUDY DESIGN:
Intervention Model Description: Participants were randomly assigned to one of three parallel groups (motivational self-talk, instructional self-talk, or control) and received the assigned intervention concurrently throughout the intervention period.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: This study employed a triple-blind design. Participants were not informed of the specific self-talk strategy being evaluated and were told only that different psychological preparation approaches were being compared. Investigators responsible for training supervision and data collection were not involved in group allocation and were blinded to intervention assignment. Outcome assessors and data analysts were blinded to group identity throughout testing and analysis. Group allocation was coded using anonymized labels until completion of all statistical analyses.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Motivational Self-Talk (Experimental): Participants in this group received a motivational self-talk intervention designed to enhance confidence, effort, and persistence during soccer training and competition.
  Interventions: Behavioral: Motivational Self-Talk Training
- Instructional Self-Talk (Experimental): Participants in this group received an instructional self-talk intervention focusing on technical execution and tactical decision-making during soccer activities.
  Interventions: Behavioral: Instructional Self-Talk Training
- Control (Experimental): Participants in the control group continued their regular soccer training without receiving any structured self-talk intervention.
  Interventions: Behavioral: No Self-Talk (Usual Training Control)

INTERVENTIONS:
Behavioral: Motivational Self-Talk Training — Participants received structured motivational self-talk training aimed at enhancing confidence, effort, and persistence during soccer training and match-related tasks. Individualized motivational cue words and phrases were developed and practiced under guidance, and participants were instructed to apply these cues consistently throughout the six-week intervention period.
  Arms: Motivational Self-Talk
Behavioral: Instructional Self-Talk Training — Participants were instructed to apply task-specific instructional self-talk cues to guide technical execution and tactical decision-making during soccer training over a six-week intervention period.
  Arms: Instructional Self-Talk
Behavioral: No Self-Talk (Usual Training Control) — Participants in the control group continued their regular soccer training and match preparation without receiving any form of structured self-talk instruction. No motivational or instructional self-talk strategies were introduced during the intervention period.
  Arms: Control

SUMMARY:
This study investigates the effects of different types of self-talk on performance and stress regulation in soccer forwards. Self-talk is a psychological technique in which athletes use specific verbal cues to guide their thoughts and actions during training and competition. Two commonly used forms are motivational self-talk, which focuses on confidence and effort, and instructional self-talk, which focuses on technical and tactical cues.

Thirty-six male soccer forwards of different competitive levels participated in this study. Players were randomly assigned to a motivational self-talk group, an instructional self-talk group, or a control group. The intervention lasted six weeks. Before and after the intervention, participants completed assessments of soccer-specific technical skills, physical performance, and match tactical behavior. Psychological measures of self-efficacy and biological indicators of stress (salivary cortisol) were also collected.

The purpose of this study is to determine whether different self-talk strategies produce different effects depending on players' competitive level and task demands. The findings are expected to provide practical guidance for the use of psychological training strategies in soccer and other team sports.

ELIGIBILITY:
Inclusion Criteria

* Male university football players aged 18-25 years
* Full-time university students regularly engaged in organized football training and competition
* At least two years of systematic football training experience
* In good general health at the time of enrollment
* No musculoskeletal injuries or medical conditions affecting football performance within the previous 6 months
* Normal or corrected-to-normal vision and hearing
* Able to understand study procedures and complete soccer-specific performance and decision-making tasks
* Provided written informed consent prior to participation

Exclusion Criteria

* History of neurological, psychiatric, or cognitive disorders that could influence decision-making or reaction time
* Current participation in structured psychological skills training programs (e.g., self-talk training, imagery, mindfulness training) outside routine football practice during the study period
* Use of medications or substances known to affect cognitive function
* Presence of any medical condition or injury contraindicating participation in football training or testing
* Failure to comply with the intervention protocol or outcome assessments

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 36 (Actual)
Dates: Start 2025-01-20 (Actual); Primary Completion 2025-03-07 (Actual); Study Completion 2025-04-05 (Actual)

PRIMARY OUTCOMES:
Match-Based Technical and Tactical Performance | Baseline and immediately after the 6-week intervention
  Match-based technical and tactical performance was assessed during regular soccer match play using standardized match analysis procedures. This outcome represents players' overall technical and tactical performance exhibited in a real match context over the intervention period.

SECONDARY OUTCOMES:
Shooting Accuracy | Baseline and immediately after the 6-week intervention
  Shooting accuracy was evaluated using a standardized soccer shooting test. Participants performed a series of shots toward predefined target zones within the goal. Shooting accuracy was calculated as the percentage of successful shots directed into the target areas, with higher percentages indicating better shooting performance.
Sport Self-Efficacy | Baseline and immediately after the 6-week intervention
  Sport self-efficacy was assessed using the Sport Self-Efficacy Scale, a validated self-report questionnaire designed to measure individuals' perceived confidence in performing sport-related skills and tasks. The scale consists of multiple items rated on a Likert-type scale, yielding a total score ranging from 10 to 50, with higher scores reflecting greater perceived self-efficacy in sport performance contexts.
Dribbling Run Performance | Baseline and immediately after the 6-week intervention
  Dribbling run performance was assessed using a standardized soccer dribbling run test. Participants completed the task while controlling the ball along a predefined running course, and performance was quantified as total completion time (seconds) recorded under standardized testing conditions.
Loughborough Soccer Passing Test Performance | Baseline and immediately after the 6-week intervention
  Passing performance was assessed using the Loughborough Soccer Passing Test (LSPT), a standardized and widely used soccer-specific passing assessment. Participants were required to complete a series of prescribed passing and ball-control actions according to the standardized test protocol. Performance was quantified as the total time (seconds) required to complete the test under controlled testing conditions.
Salivary Cortisol Concentration | Baseline and immediately after the 6-week intervention
  Salivary cortisol concentration was assessed as an index of physiological stress response. Saliva samples were collected using standardized saliva collection procedures and cortisol levels were quantified using enzyme-linked immunosorbent assay (ELISA) methods under controlled laboratory conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Sport University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No
Individual participant data will not be shared due to participant confidentiality and institutional data protection policies.